CLINICAL TRIAL: NCT04311645
Title: Role of Oral Activated Charcoal in Decreasing Blood Urea, Creatinine and Phosphorous in Chronic Kidney Disease
Brief Title: Role of Activated Charcoal in Decreasing Blood Urea, Creatinine and Phosphorous
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Farrag Sayed Mohamed, Resident Doctor, internal medicine department, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Charcoal CKD progression
Record Dates: First submitted 2020-03-14; First posted 2020-03-17 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Chronic Kidney Disease stage3
MeSH Terms: interventions — Charcoal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1st group (Other): Oral activated charcoal in a dose of 30 gm/day
  Interventions: Drug: Activated charcoal
- 2nd group (Other): Dry seeds in a dose of 1 gm/ day
  Interventions: Dietary Supplement: Dry seeds
- 3rd group (No Intervention): control group

INTERVENTIONS:
Drug: Activated charcoal — Activated charcoal
  Arms: 1st group
Dietary Supplement: Dry seeds — Dry seeds
  Arms: 2nd group

SUMMARY:
The study aims to explore the ability of Oral activated charcoal to adsorb uremic toxins limiting the progression of chronic kidney disease and delaying the need for hemodialysis in patients with CKD stages III and IV.

To compare its effect with the effect of dry seeds as absorbents of uremic toxins

DETAILED DESCRIPTION:
In recent years, chronic kidney disease(CKD) has become a worldwide public health issue.

The main factors affecting the prognosis of patients with chronic kidney disease are its complications, including cardiovascular and cerebrovascular diseases, malnutrition, inflammation, atherosclerosis syndrome, and anemia.

The accumulation of uremic toxins, such as indoxyl sulfate and p-cresyl sulfate, is implicated in the progression of renal failure and cardiovascular disease.

For many patients, chronic kidney disease (CKD) is a progressive condition marked by deteriorating renal function ultimately leading to end-stage renal disease (ESRD) and many patients refuse to start chronic hemodialysis.

Therapeutic approaches that decrease the level of uremic toxins are a rational method for inhibiting this progression.

Many researches have been done aiming to find alternatives for chronic hemodialysis either for economic issues or psychological issues especially in elderly patients, as example:

* Gum Arabic in the remedy and amelioration of kidney dysfunction and end-stage renal disease
* skin as excretory root for urea, increasing sweat from sweat glands can support kidney function by excreting a good amount of what kidneys naturally excrete.
* The oral charcoal adsorbent reduces serum levels of indoxyl sulfate through adsorption of indole converted from dietary tryptophan in the gastrointestinal tract decreasing serum creatinine and urea level .

In this study, the clinical data supporting the role of oral activated charcoal in a dose of 30gm/ day for slowing the progression of CKD will be reviewed.

In this study, a trial will be done using dry seeds (lentils as an example) as an absorbent for uremic toxins comparing its effect with the effect of oral activated charcoal.

ELIGIBILITY:
Inclusion Criteria:

Patients with CKD stages iii and iv

Patients with age more than 18 years old

Exclusion Criteria:

Patients on regular hemodialysis

Patients with age less than 18 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Mean of blood urea, creatinine and phosphorous in patients with CKD before and after oral activated charcoal | baseline
  to asses the mean of blood urea, creatinine and phosphorous in CKD patient before and after administration of activated charcoal

SECONDARY OUTCOMES:
comparison of dry seeds and activated charcoal in limitting progression of chronic kidney disease | baseline
  To compare dry seeds with activated charcoal as as alternative natural cheap methods that may help in limitting progression of CKD by measuring blood urea, creatinine, and phosphorous in all 3 groups of the study

REFERENCES:
- [Background] Brunori G, Viola BF, Maiorca P, Cancarini G. How to manage elderly patients with chronic renal failure: conservative management versus dialysis. Blood Purif. 2008;26(1):36-40. doi: 10.1159/000110561. Epub 2008 Jan 10. PMID 18182793
- [Background] Niwa T. Indoxyl sulfate is a nephro-vascular toxin. J Ren Nutr. 2010 Sep;20(5 Suppl):S2-6. doi: 10.1053/j.jrn.2010.05.002. PMID 20797565
- [Background] Niwa T, Emoto Y, Maeda K, Uehara Y, Yamada N, Shibata M. Oral sorbent suppresses accumulation of albumin-bound indoxyl sulphate in serum of haemodialysis patients. Nephrol Dial Transplant. 1991;6(2):105-9. doi: 10.1093/ndt/6.2.105. PMID 1906999
- [Background] Xie L, Jin L, Feng J, Lv J. The Expression of AQP5 and UTs in the Sweat Glands of Uremic Patients. Biomed Res Int. 2017;2017:8629783. doi: 10.1155/2017/8629783. Epub 2017 Nov 27. PMID 29279852
- [Background] Blacher J, Guerin AP, Pannier B, Marchais SJ, London GM. Arterial calcifications, arterial stiffness, and cardiovascular risk in end-stage renal disease. Hypertension. 2001 Oct;38(4):938-42. doi: 10.1161/hy1001.096358. PMID 11641313
- [Background] Mizobuchi M, Towler D, Slatopolsky E. Vascular calcification: the killer of patients with chronic kidney disease. J Am Soc Nephrol. 2009 Jul;20(7):1453-64. doi: 10.1681/ASN.2008070692. Epub 2009 May 28. PMID 19478096
- [Background] Cook WL, Jassal SV. Prevalence of falls among seniors maintained on hemodialysis. Int Urol Nephrol. 2005;37(3):649-52. doi: 10.1007/s11255-005-0396-9. PMID 16307356
- [Background] Kurella M, Covinsky KE, Collins AJ, Chertow GM. Octogenarians and nonagenarians starting dialysis in the United States. Ann Intern Med. 2007 Feb 6;146(3):177-83. doi: 10.7326/0003-4819-146-3-200702060-00006. PMID 17283348
- [Background] Friedman EA. Bowel as a kidney substitute in renal failure. Am J Kidney Dis. 1996 Dec;28(6):943-50. doi: 10.1016/s0272-6386(96)90399-6. PMID 8957051